CLINICAL TRIAL: NCT07275255
Title: Non-Specific Chronic Low Back Pain: Investigation of Interoceptive Awareness, Physical Activity Level, Body Awareness and Emotional Status in Individuals With Non-Specific Chronic Low Back Pain
Brief Title: Interoceptive Awareness, Physical Activity, Body Awareness and Emotional Status in Individuals With Non-Specific Chronic Low Back Pain
Acronym: NSCLBP-AWARE
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Other Study IDs: ISTINYE-PT-NSCLBP-2025
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Lower Back Pain Chronic; Non Specific Chronic Low Back Pain
Keywords: Interoceptive Awareness; Body Awareness; Non-specific Chronic Low Back Pain; Chronic Low Back Pain; Alexithymia; Physical Activity
MeSH Terms: conditions — Affective Symptoms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-specific Chronic Low Back Pain Group: A cohort of adults aged 18-65 diagnosed with non-specific chronic low back pain. Participants will complete validated self-report questionnaires assessing interoceptive awareness, body awareness, emotional status, physical activity level, and pain intensity.

SUMMARY:
This observational cross-sectional study aims to examine the relationships between interoceptive awareness, physical activity level, body awareness, emotional status, and pain intensity in individuals with non-specific chronic low back pain. Non-specific chronic low back pain refers to pain in the lumbar region lasting for at least three months without an identifiable structural or pathological cause.

Participants aged 18-65 years who meet the diagnostic criteria for non-specific chronic low back pain will be evaluated using validated self-report questionnaires. These include measures of interoceptive awareness, body awareness, alexithymia, physical activity level, and pain intensity. Sociodemographic and clinical characteristics such as age, gender, education level, duration of pain, medication use, height, weight, and BMI will also be collected.

The purpose of the study is to better understand how internal body perception, physical activity, emotional processing, and body awareness interact with pain experience in this population. Findings may contribute to the development of individualized rehabilitation programs and inform clinicians about the multidimensional factors influencing chronic low back pain.

DETAILED DESCRIPTION:
This study is designed as a quantitative, cross-sectional, observational investigation involving adults aged 18-65 years diagnosed with non-specific chronic low back pain (ns-cLBP). Non-specific chronic low back pain is defined as lumbar pain lasting at least three months without an identifiable structural pathology such as tumor, infection, fracture, inflammatory disease, spinal stenosis, or radiculopathy. Chronic low back pain is known to negatively affect daily activities, emotional well-being, physical function, and quality of life. Recent literature suggests that interoceptive awareness, emotional regulation, body awareness, and physical activity level play important roles in the pain experience and coping mechanisms of individuals with chronic pain.

Despite growing evidence, the multidimensional relationships among interoceptive awareness, body awareness, physical activity level, emotional status, and pain severity have not been comprehensively examined in individuals with non-specific chronic low back pain. Therefore, this study aims to fill this gap by evaluating these variables together.

A total of approximately 130 participants will be recruited. Sociodemographic and clinical data including age, gender, marital status, education level, duration of pain, medication use, smoking status, height, weight, BMI, and waist-to-hip ratio will be recorded. The following validated self-report questionnaires will be administered:

Interoceptive awareness: Multidimensional Assessment of Interoceptive Awareness (MAIA/MAIA-2)

Body awareness: Body Awareness Rating Questionnaire - Turkish (BARQ-T)

Emotional status (alexithymia): Toronto Alexithymia Scale-20 (TAS-20)

Pain intensity: Visual Analog Scale (VAS)

Physical activity level: International Physical Activity Questionnaire - Short Form (IPAQ-SF)

Data analysis will be performed using SPSS (v.27). Normality will be assessed with the Shapiro-Wilk test. Parametric or non-parametric correlation tests (Pearson or Spearman) will be used to examine relationships between variables. Group comparisons (e.g., sex, age groups, physical activity levels) will be conducted using independent samples t-tests or Mann-Whitney U tests depending on data distribution. Statistical significance will be set at p < 0.05.

The study is expected to contribute new insights into the emotional, cognitive, and sensory mechanisms underlying chronic low back pain. Understanding these multidimensional interactions may help clinicians develop more targeted and individualized rehabilitation strategies, particularly those incorporating body awareness and interoception-based therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Diagnosed with non-specific chronic low back pain.
* Duration of pain ≥ 3 months.
* Self-reported average pain score ≥ 4/10 on the Visual Analog Scale.
* Ability to understand and complete self-report questionnaires.

Exclusion Criteria:

* Low back pain due to specific pathologies (e.g., tumor, infection, fracture, inflammatory disease).
* Serious systemic, neurological, or psychiatric comorbidities.
* History of spinal surgery within the past year.
* Pregnancy.
* Language or cognitive impairments preventing questionnaire completion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-65 years diagnosed with non-specific chronic low back pain for at least 3 months. Participants will be recruited from the physiotherapy and rehabilitation outpatient clinic (Fizyotem) at Istinye University. Individuals must be able to understand and complete self-report questionnaires. A total of approximately 130 participants are expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Interoceptive Awareness Score (MAIA/MAIA-2) | Baseline
  Interoceptive awareness will be assessed using the Multidimensional Assessment of Interoceptive Awareness (MAIA/MAIA-2). The scale consists of 37 items rated on a 5-point Likert scale, yielding scores for eight subscales. Higher scores indicate greater interoceptive awareness.

SECONDARY OUTCOMES:
Body Awareness Score (BARQ-T) | Baseline
  Body awareness will be measured using the Body Awareness Rating Questionnaire - Turkish (BARQ-T). The scale assesses perception of bodily sensations and awareness-related behaviors. Higher scores indicate greater body awareness.
Alexithymia Score (Toronto Alexithymia Scale-20) | Baseline
  Emotional status will be assessed using the Toronto Alexithymia Scale-20 (TAS-20), a 20-item questionnaire measuring difficulty identifying feelings, difficulty describing feelings, and externally oriented thinking. Higher scores represent higher levels of alexithymia.
Physical Activity Level (IPAQ-SF) | Baseline
  Physical activity will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). Total activity will be calculated in MET-minutes/week, and participants will be categorized as low, moderate, or high activity level.

OTHER OUTCOMES:
Pain Intensity Score (Visual Analog Scale) | Baseline
  Pain intensity will be measured using a 10-cm Visual Analog Scale (VAS), where 0 represents "no pain" and 10 represents "worst imaginable pain." Scores are recorded in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Gül Deniz Yılmaz Yelvar, Assoc. Prof., Study Chair — Istinye University, Institute of Graduate Studies, Department of Physiotherapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality considerations.